CLINICAL TRIAL: NCT03306758
Title: The Efficiency and Safety of Sodium Bicarbonate on Uric Acid in Patients With Asymptomatic Hyperuricemia or Gout
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Jiang lindi, Chief, Professor, Department of Rheumatology, Shanghai Zhongshan Hospital, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2017-136R
Record Dates: First submitted 2017-09-27; First posted 2017-10-11 (Actual); Last update posted 2017-10-11 (Actual); Status verified 2017-09

CONDITIONS: Asymptomatic Hyperuricemia; Gout
MeSH Terms: conditions — Gout | interventions — Sodium Bicarbonate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: sodium bicarbonate (Experimental)
  Interventions: Drug: Sodium Bicarbonate
- No Intervention (No Intervention)

INTERVENTIONS:
Drug: Sodium Bicarbonate — Sodium Bicarbonate was given 1g tid for one month
  Arms: Experimental: sodium bicarbonate

SUMMARY:
This study evaluate the serum uric acid lowering effect of sodium bicarbonate as well as its safety in patients with asymptomatic hyperuricemia or gout. Half of the participants will receive sodium bicarbonate only, while the other half receive none.

ELIGIBILITY:
Inclusion Criteria:

1. Sign informed consent form;
2. Serum uric acid ≥420mmol/L;
3. Within the age range of 18-65 years old;
4. Within the BMI range of 18-30kg/m2;
5. Both men and women are eligible

Exclusion Criteria:

1. General situations

   * Pregnancy or lactation；
   * Participants who can't take contraception during the study or within one month after the completion of the intervention;
   * Situations which will harm the participants;
   * Participants with bad compliance.
2. Taking part in another trail
3. Gout flares happening over the last one month;
4. Administration of medications over the last one month, including: allopurinol, Febuxostat,benzbromarone, and/or sodium bicarbonate；
5. urine pH>7.0;
6. Hepatic function：ALT and/or AST and/or TB>1.5 upper limit of normal (ULN);
7. Renal function：eGFR<60 ml/min for MDRD and/or urine protein>0.5g/24h；
8. Hypertension：>140/90mmHg;
9. Type 2 diabetes or taking drugs for lowering glucose (not including prediabetes);
10. Urinary stone,urinary infection;
11. Taking drugs ove the last one month and during the trial, including：thiazide diuretic, Loop diuretics, pyrazinamide,ethambutol, tacrolimus, niacin, aspirin, estrogen, losartan, amlodipine, reserpine, vitamin C，fenofibrate，atorvastatin， sulfonylureas，biguanides，NSAIDs;
12. Disease which influence serum uric acid, such as cancer, lymphoma, and etc.
13. Severe disorders involving heart, liver, kidneys, brain, lungs,digestive tract, rheumatoid disease, blood, endocrine, infection, and etc;
14. Blood donation or excessive loss of blood over the last 3 month.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2018-07-31 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Serum uric acid | 1 month after randomization
  Change from baseline serum levels of uric acid at 1 month

SECONDARY OUTCOMES:
Fraction excretion of uric acid | 1 month after randomization
  Change from baseline fraction excretion of uric acid at 1 month